CLINICAL TRIAL: NCT04382001
Title: Further Investigations of Heart Rate Variability During the Menstrual Cycle
Brief Title: Heart Rate Variability During the Menstrual Cycle
Status: Completed | Type: Observational
Sponsor: SPD Development Company Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: PROTOCOL-1196
Record Dates: First submitted 2020-05-06; First posted 2020-05-11 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Ovulation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, women will be required to wear a chest heart rate monitor and wrist heart rate monitor daily and collect daily early morning urine samples for the duration of one complete menstrual cycle. This will enable comparisons between data collected from the heart rate monitor and hormone analysis in urine samples to be made.

DETAILED DESCRIPTION:
This study is a prospective observational study of women's heart rate and heart rate variability throughout one complete menstrual cycle. A minimum of 10 volunteers aged 18 years of age or over will be recruited via a variety of methods according to the criteria detailed in section 9. They will be required to wear a chest heart rate monitor and wrist heart rate monitor for 1 hour each day, and throughout the night for one menstrual cycle. In addition, a daily early morning urine sample will be collected throughout the study.

Urine samples will be returned to SPD on a regular basis for measurement of urinary hormones related to pregnancy and fertility. Data collected via the monitors including heart rate and heart rate variability will be downloaded for comparison.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years of age and over
* Regular menstrual cycles (23-35 days in length)-

Exclusion Criteria:

* Taking any hormonal medications
* Taking any medications that may affect heart rate
* Known heart condition or use of a pacemaker
* Skin condition where there is sensitivity to wearing a skin monitor
* Currently suffering with anxiety or panic attacks
* Pregnant or breastfeeding
* Undertaking any frequent travel or long-haul flights during the course of the study
* Does not have access to an Apple iPhone or iPad with Bluetooth 4.0 (or later) and iOS 10.0 (or later)

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Adult female
Study Population: Healthy volunteers
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-05-06 (Actual); Study Completion 2021-05-06 (Actual)

PRIMARY OUTCOMES:
Heart rate | 1 month
  Heart rate at time points throughout the menstrual cycle
Heart Rate | 1 month
  Heart rate variability at time points throughout the menstrual cycle
Day of Ovulation | 1 month
  Day of ovulation determined by urinary LH surge +1 day
Fertile Window | 1 month
  Fertile window onset determined by E3G surge
Fertile window | 1 month
  Fertile window closure determined by P3G rise

SECONDARY OUTCOMES:
Comparisons between wrist and chest band monitors | 1 month
  Agreement between wrist band and chest band heart rate data

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Johnson, Study Director — SPD Development Company
Locations (1):
- SPD Development Company Ltd, Bedford, Bedfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided